CLINICAL TRIAL: NCT00006460
Title: A Phase I/II Trial of Conformal Radiotherapy and Hyperbaric Oxygen for Patients With Newly Diagnosed Glioblastoma
Brief Title: Radiation Therapy Plus Hyperbaric Oxygen in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barrett Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068256; UCMC-00021401; NCI-V00-1626
Record Dates: First submitted 2000-11-06; First posted 2004-02-03 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2002-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Hyperbaric Oxygenation; Radiotherapy

INTERVENTIONS:
Drug: hyperbaric oxygen
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Hyperbaric oxygen may increase the effectiveness of radiation therapy. Combining hyperbaric oxygen with radiation therapy may be an effective treatment for glioblastoma multiforme.

PURPOSE: Phase I/II trial to study the effectiveness of combining radiation therapy with hyperbaric oxygen in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility and toxicity of hyperbaric oxygen combined with conformal radiotherapy in patients with newly diagnosed glioblastoma multiforme. II. Determine the efficacy of this regimen in terms of radiographic tumor response, time to tumor progression, and survival in these patients.

OUTLINE: Within 2 weeks after surgery, patients receive hyperbaric oxygen over 90 minutes once daily, followed by conformal radiotherapy twice daily 5 days a week for 17 days in the absence of unacceptable toxicity. Patients are followed within 2 weeks and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 5-10 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven newly diagnosed glioblastoma multiforme Measurable residual tumor by MRI after biopsy or craniotomy

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 70-100% Life expectancy: More than 8 weeks Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Pulmonary: No severe pulmonary disease (e.g., emphysema with carbon dioxide retention) No untreated pneumothorax Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other malignancy within the past 5 years except epithelial skin cancer No psychological, familial, sociological, or geographical conditions that would preclude study No intractable seizure disorder

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior or concurrent bleomycin Endocrine therapy: Not specified Radiotherapy: No prior cranial radiotherapy Surgery: See Disease Characteristics Other: No other prior therapy, including adjuvant therapy, for glioblastoma multiforme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E. Warnick, MD, Study Chair — Barrett Cancer Center
Locations (1):
- Barrett Cancer Center, The University Hospital, Cincinnati, Ohio, United States